CLINICAL TRIAL: NCT01347502
Title: Bacterial Contamination of Smart Phones of Health Care Workers
Brief Title: Prevalence of Bacterial Contamination on Smart Cell Phone vs. Non-smart Phone
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jae-Joon Yim, professor, Seoul National University Hospital
Other Study IDs: smartphone_SNU
Record Dates: First submitted 2011-05-03; First posted 2011-05-04 (Estimated); Last update posted 2012-07-09 (Estimated); Status verified 2012-07

CONDITIONS: Health Care Workers, Including Physicians, Nurses, and Nursing Aids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HCPs with smartphone: healthcare providers in MICU who have smart cellular phones
- HCP with non-smart phones: healthcare providers in MICU who have non-smart cellular phones

SUMMARY:
Using smartphone is increasing in hospital with various purpose and it has more extended surface than non-smart phone. Therefore investigators can consider the bacterial contamination rate of smartphone will be higher than that of non-smartphone.

DETAILED DESCRIPTION:
Hospital-acquired infections(HAI) are causing grave concern in almost all the hospitals of the world and causing increased morbidity and mortalities.

The transmission of HAI occurs through hospital staff and inanimate hospital environment, equipment, and devices that the hospital staff use.Recently, cellphones (CP) were blamed to cause nosocomial infections.

The mobile phones are used routinely all day long but not cleaned properly, as health care workers' may do not wash their hands as often as they should. The aim of the present study was to evaluate the prevalence of bacterial contamination of mobile phones in ICU health care providers. and especially compare the contamination rate between smartphone and non-smartphone.

Using smartphone is increasing in hospital with various purpose and it has more extended surface than non-smart phone. therefore we can consider the bacterial contamination rate of smartphone will be higher than that of non-smartphone.

ELIGIBILITY:
Inclusion Criteria:

* healthcare providers of MICU who have cellular phones

Exclusion Criteria:

* healthcare providers of MICU who have not cellular phones

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthcare providers of MICU in Seoul national university hospital and Seoul national university Bundang hospital who have cellular phones
Sampling Method: Non-Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2011-04; Primary Completion 2011-06 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Joon Yim, MD, Principal Investigator — Seoul National University Hospital
Locations (3):
- South Korea (3):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul Metropolitan Government Seoul National University Boramae Medical Center, Seoul
  - Seoul National University Hospital, Seoul

REFERENCES:
- [Derived] Lee YJ, Yoo CG, Lee CT, Chung HS, Kim YW, Han SK, Yim JJ. Contamination rates between smart cell phones and non-smart cell phones of healthcare workers. J Hosp Med. 2013 Mar;8(3):144-7. doi: 10.1002/jhm.2011. Epub 2013 Feb 15. PMID 23418134